CLINICAL TRIAL: NCT07279701
Title: The Effect of Near-infrared Spectroscopy on the Success of Peripheral Venous Access: a Pilot Randomized Controlled Study
Brief Title: The Effect of Near-infrared Spectroscopy on the Success of Peripheral Venous Access
Acronym: PEDVEIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, prof. MD, PhD, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PEDVEIN
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Intravenous Cannulation
Keywords: pediatric; near-infrared imaging; periferal vein cannulation; difficult intravenous access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- VeinViewer Flex (Experimental): The periferal vein cannulation will be aided by concurrent near-infrared imaging by device VeinViewer Flex using AVIN™ (Active Vascular Imaging Navigation).
  Interventions: Device: Use of near-infrared imaging by VeinViewer Flex of periferal veins
- Landmark (No Intervention): The peripheral vein cannulatoon will be provided by usual landmark technique, without any other imaging device.

INTERVENTIONS:
Device: Use of near-infrared imaging by VeinViewer Flex of periferal veins — The projected near-infrared light is absorbed by the blood and reflected by surrounding tissue, captured, processed, and digitally projected in real time directly onto the skin surface. It provides an accurate, real-time image of the patient's blood pattern.
  Patented VeinViewer technology using AVIN™ (Active Vascular Imaging Navigation) allows the blood vessels to be seen down to a depth of 10 mm. With VeinViewer, physicians can see peripheral veins, bifurcations, and valves and assess venous filling/flushing in real time.
  Arms: VeinViewer Flex

SUMMARY:
The goal of this clinical trial is to learn if using near-infrared imaging in pediatric vein cannulation is leading to higher success rate. The main question it aims to answer is:

is there higher success of first attempt in periferal vein cannulation? does it lower overall number of attempts to successful cannulation?

DETAILED DESCRIPTION:
Providing venous access in pediatric anesthesia and intensive care is among the basic and necessary interventions for blood sampling and administration of drugs and possibly transfusion products and derivatives.

In anesthesia, effective provision of venous access is a prerequisite for safe anesthesia. In pediatric patients and newborns, provision of venous access is complicated by patient non-cooperation, but primarily by the smaller diameter of the vessels and often limited possibility of direct visualization, or limited possibility of palpation of the vessel under visual control. Ultrasound is currently used to facilitate provision of IV access, however, imaging under the USG probe and its subsequent puncture requires high skill of medical personnel and is preferentially applied by medical staff in the conditions of the Czech Republic. Near-infrared imaging (IR) allows direct visualization of superficial vascular bed and may potentially be associated with higher puncture success rates (higher first attempt success, reduction of total attempts).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients admitted to the inpatient section of the Department of Pediatric Anesthesiology and Resuscitation, Brno University Hospital
* Pediatric patients in the anesthesia section of the Department of Pediatric Anesthesiology and Resuscitation, Brno University Hospital
* Indicated insertion of peripheral venous access
* Consent of the patient/legal representative to the study

Exclusion Criteria:

* Disagreement with the study
* Not indicated insertion of peripheral venous access (according to clinical condition and decision of the attending physician)
* A device for near-infrared imaging of the venous bed is not available

Ages: 0 Days to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of first attempt in peripheral vein cannulation | Periprocedural
  Success rate of first attempt in periferal vein cannulation
Number of attempts | Periprocedural
  Overall number of attempts needed to secure periferal vein access

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof, MD, PhD, Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided